CLINICAL TRIAL: NCT03620513
Title: Pretreatment With Topical Anesthesia or Decongestant for Reducing Pain and Discomfort During Fiberoptic Nasal Pharyngoscopy and Laryngoscopy: A Double Blind Randomized Study
Brief Title: Pretreatment to Reduce Pain and Discomfort During Fiberoptic Nasal Pharyngoscopy and Laryngoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lumbini Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 142
Record Dates: First submitted 2018-07-08; First posted 2018-08-08 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Throat Disorder
MeSH Terms: interventions — Nasal Decongestants; Anesthesia; Oxymetazoline; Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Four arms of study group with equal number of subjects in each group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal Saline nasal spray (Placebo Comparator): Two spray (via atomizer) of normal saline in each nostril five minutes prior to fiberoptic procedure
  Interventions: Drug: Normal saline
- Decongestant (Oxymetazoline 0.05%) (Experimental): Two sprays via atomizer (about 0.18 ml) of oxymetazoline 0.05% (Nasivion) in each nasal cavity five minutes prior to fiberoptic procedure. Two sprays will be given at the gap of ten seconds.
  Interventions: Drug: Decongestant (oxymetazoline 0.05%)
- Anesthesia (lidocaine 15%, Nummit) (Experimental): Two sprays of 15% lidocaine (Nummit) will be give in each nasal cavity five minutes prior to fiber optic procedure. Two sprays will be given at the gap of ten seconds.
  Interventions: Drug: Anesthesia (Lidocaine 15%)
- Decongestant and Anesthesia (Experimental): In this group decongestants and anesthesia (oxymetazoline and lidocaine) sprays will be used. Decongestant (Oxymetazoline 0.05%) will be give as described above. After two minutes, lidocaine 15% (Nummit) spray will be given as described above. Procedure will be done after five minutes of decongestant.
  Interventions: Drug: Decongestants and Anesthesia (oxymetazoline and lidocaine)

INTERVENTIONS:
Drug: Decongestant (oxymetazoline 0.05%) — As described in arm/group
  Other Names: Nasivion
  Arms: Decongestant (Oxymetazoline 0.05%)
Drug: Anesthesia (Lidocaine 15%) — As described in arm/group
  Other Names: Nummit
  Arms: Anesthesia (lidocaine 15%, Nummit)
Drug: Decongestants and Anesthesia (oxymetazoline and lidocaine) — As described in arm/group
  Other Names: Nasivion and Nummit
  Arms: Decongestant and Anesthesia
Drug: Normal saline — Spray of normal saline as premedication
  Arms: Normal Saline nasal spray

SUMMARY:
Fiberoptic laryngoscopy (FOL) is one of the most common procedure done in an Ear Nose Throat (ENT) clinic. Topical anesthesia or decongestant or both have been used to improve patient comfort level during the procedure. Recently, role of these agents has been questioned. The investigators would like to study whether topical anesthesia or decongestant or their combination provide any benefit to the patients undergoing FOL.

DETAILED DESCRIPTION:
Patient undergoing Fiberoptic laryngoscopy (FOL) will be randomized into four groups by block randomization. Group one will receive atomized spray of normal saline as placebo before the procedure. Group two will receive two sprays of atomized oxymetazoline (approx 0.18 ml of 0.05% oxymetazoline) with a gap of 10 seconds in between the sprays. Group three will receive two sprays of 15% lidocaine with a gap of 10 seconds in between the sprays. Group four will receive two sprays of oxymetazoline and then two sprays of lidocaine at an interval of two minutes.

Sample size calculation: With alpha error of 0.05, power of .8, mean discomfort scale for placebo of 2.8 (literature review) and SD of 1.1, presuming that the treatment would be able to reduce discomfort by at least 25%, with two tailed test and same SD, minimum sample size would be 40 in each group.

To reduce bias, all the procedure will be performed by senior consultants. Patients and the person performing the procedure will be blinded.

Discomfort of pre-medication, discomfort of scope insertion, pain due to scope insertion, and ease of procedure will be scored as VAS score (1 to 10, 1 is least and 10 is most). Also, patient will be asked how likely s/he is to recommend the similar procedure to his/her friends and family members in case they need to undergo the same. Side effects of pre-medication and procedure will also be noted.

Outcome variables among the groups will be compared using ANOVA test if they are normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fiberoptic naso pharyngo laryngoscopy in OPD setting
* Consent to study
* above 18 years

Exclusion Criteria:

* gross nasal mass
* pregnants
* known hypersensitivity to the drugs used for premedication
* who cannot respond to questionnaire during data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Discomfort of procedure (fiberoptic nasopharyngolaryngoscopy) as VAS 1-10 | At the end of the procedure
  Discomfort will be scored as VAS on a scale of 1 to 10 (1 is least, 10 is most)

SECONDARY OUTCOMES:
Discomfort of pre-treatment as VAS 1-10 | four minutes from the first spray
  Discomfort will be scored as VAS on a scale of 1 to 10 (1 is least, 10 is most)
Prevalence of adverse effects of pre-medication | four minutes from the first spray
  allergy, burning pain, altered taste, chocking sensation, headache will be asked and recorded
Pain due to procedure as VAS 1-10 | At the end of the procedure
  Pain will be scored as VAS on a scale of 1 to 10 (1 is least, 10 is most)
Ease of procedure as VAS 1-10 | At the end of the procedure
  Ease will be scored as VAS on a scale of 1 to 10 (1 is least, 10 is most)
Prevalence of adverse effects of procedure | At the end of the procedure
  bleeding, gag, nausea, vomiting will be noted
Likely to recommend (not likely, can not say, very likely) | At the end of the procedure
  Patient will be asked, "How likely you are to recommend this procedure to your relative in case they are advised to". It will be scored as 1-Not at all; 2-not sure; 3-Strongly recommend

CONTACTS AND LOCATIONS:
Overall Officials: Anup Acharya, MS, Principal Investigator — Associate Professor
Locations (1):
- Lumbini Medical College, Tānsen, Palpa, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data via journal website or on request to the researcher
Supporting Information: SAP, Analytic Code
Time Frame: As soon as article is published online. It will be available for good.